CLINICAL TRIAL: NCT00507351
Title: Ambulatory Cancer Pain Management: A Feasibility Study
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0841
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer
Keywords: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer; Pain Management; Questionnaire; Survey
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Agnosia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer Pain Management: Patients receiving chemotherapy for breast, colon, lung, or prostate cancer.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 3 questionnaires that will take 20 minutes total to complete.
  Other Names: Survey

SUMMARY:
The primary purpose of this study is to examine the feasibility of collecting pain and other symptom data in outpatient treatment centers across multiple institutions in the Texas Medical Center (TMC). We will also examine the prevalence and severity of cancer-related pain and begin to identify other commonly reported symptoms in outpatient settings. Factors that interfere with management of pain will also be examined. Additionally, the study will explore patient satisfaction with pain management and pain education in outpatient settings. The specific aims of this study include:

Primary Objective:

-Explore the feasibility of a collaborative effort by oncology nurses to collect pain and symptom data across multiple institutions that care for ambulatory cancer patients in the TMC.

Secondary Objectives:

* Describe the prevalence and severity of pain and other symptoms in persons with breast, colorectal, lung, or prostate cancer who are receiving chemotherapy in the outpatient setting.
* Describe factors that interfere with adequate pain management in these patients.
* Examine patient satisfaction with pain management and patient education about pain management.

DETAILED DESCRIPTION:
You will be asked to complete 3 questionnaires that will take a total of about 20 minutes to complete. Your name or medical record number will not appear on the questionnaires. You will be assigned a study subject code number. The study chair will keep a file that links your name to the code.

The first questionnaire will ask for basic demographic information (such as gender, ethnicity, and education) and your current chemotherapy and pain medications. If you cannot remember the names of these medications, researchers will locate them in your M. D. Anderson medical record.

The second questionnaire asks you to rate your pain and a variety of symptoms (for example, fatigue and nausea).

The last questionnaire includes 3 sections. The first section asks about your beliefs about pain and its treatment. The second part asks for your opinion about your pain management and about the education you have received about pain management. On the last page, you will be asked to use a picture of the outline of a body to show the researchers where you have pain.

Once you have completed these questionnaires, you will be considered off-study.

This is an investigational study. Up to 125 patients will take part in this study. Up to 35 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of breast, colorectal, lung, or prostate cancer (any histological type).
2. Currently undergoing chemotherapy.
3. Age 18 or older.
4. Able to read, write, and speak English.
5. Able to understand the purpose of this study.
6. Must be a patient at one of the four participating institutions.
7. Must be receiving the 2nd, 3rd, or 4th cycle of chemotherapy.

Exclusion Criteria:

1. Receiving chemotherapy in preparation for a bone marrow or stem cell transplant
2. Received a bone marrow or stem cell transplant
3. Age 17 or younger
4. Receiving weekly chemotherapy.
5. Receiving hormonal therapy alone.
6. Receiving radiation or chemoradiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy for breast, colon, lung, or prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pain and symptom data across multiple institutions | Survey data collection taking 30 minutes, collecation accomplished at multiple sites over 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anita Broxson, RN, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Memorial Hermann Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Michael E. DeBakey Veterans Administration Medical Center, Houston, Texas
  - U.T.M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org